CLINICAL TRIAL: NCT05078645
Title: Improving Sleep and Reducing External Stimuli With the Maya: a Pilot Study on Experience, Feasibility and Applicability
Brief Title: Improving Sleep and Reducing External Stimuli With the Maya
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Bram Tilburgs, Principal Investigator, Radboud University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-13078
Record Dates: First submitted 2021-09-13; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Pilot study with a crossover design. Half of the patients will use the Maya on the first, third and fifth day of their admission and will not use the maya on the second fourth and sixth day (group 1). The other half will use the Maya on the second, fourth and sixth day of their admission and will not use the maya on the first, third and fifth day (group 2). Group allocation will be randomised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Maya use on 1st, 3th and 5th day (Other): Group 1 uses the Maya on the 1st, 3th and 5th day and not on the 2nd, 4th and 6th day of their admission to either the ICU, MC or CCU.
  Interventions: Device: Maya
- Group 2: Maya use on the 2nd, 4th, and 6th day (Other): Group 2 uses the Maya on the 2nd, 4th and 6th day and not on the 1st, 3th, and 5th day of their admission to either the ICU, MC or CCU.
  Interventions: Device: Maya

INTERVENTIONS:
Device: Maya — The Maya is a cover which can be placed over the end of the patients bed. The Maya aims to reduce light and sound nuisances and enhance patients' privacy

SUMMARY:
Lack of sleep is a large problem for many patients in hospitals. Common causes are nuisances by light and sound. Especially with critically ill patients in the Intensive Care unit (ICU), Medium Care Unit (MCU) and Cardiac Care Unit (CCU), who are are monitored intensively, a lack of sleep often occurs.

Patients with a lack of sleep more offer suffer from delirium, are more often anxious and stressed, and have a longer length of stay in the hospital. Also, patients' lack of sleep enhances nurses workloads during nightshifts. Because of this, there is a strong need for innovative devices which aim to limit the light and sound nuisances and thereby enhance patients' quality of sleep in the ICU, MC and CCU.

The Maya is a special "cover" which can be placed over the head of the bed. As a result patients are able to limit light and sound nuisances and enhance their privacy.

With this pilot-study we aim to determine:

* The feasibility and experiences of patients and healthcare professionals with the Maya.
* To determine the effect size of dependent variables which can be used in future studies.

ELIGIBILITY:
Inclusion Criteria:

* adult ICU, MC or CCU patients with 5 to 7 expected number of admission days
* patients with an expected Richmond Agitation Sedation Scale (RASS) of >-3 and < +3
* patients who speak Dutch (because of the qualitative evaluation of the Maya)

Exclusion Criteria:

* patients with severe brain damage
* patients with a severe psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Quality of sleep | up to six days
  patients' quality of sleep is measured once a day with the Richard Campbell Sleep Questionnaire (RCSQ); (minimum score 0 = worst sleep - maximum score 100 = best sleep)

SECONDARY OUTCOMES:
NRS sleep | up to six days
  Patients' sleep is measured once a day with the sleep numeric rating scale (NRS sleep); (minimum score 0 = worst sleep - maximum score 10 = best sleep)
Anxiety | up to six days
  Patients' anxiety is measured once a day with the Daily Assesment of symptoms of Anxiety (DAS-A); (minimum score 0 = no anxiety - maximum score 24 = a lot of anxiety)
NRS Stress | up to six days
  Patients' stress is measured once a day with the stress numeric rating scale (NRS-stress); (minimum score 0 = no stress - maximum score 10 = most imaginable stress)
Arousal | up to six days
  patients' arousal is measured once a day with the Richmond Agitation Sedation Scale (RASS); (minimum score -5 = no reaction - maximum score = 4 very agitated)
Delirium CCU | up to six days
  CCU patients' delirium is measured once a day with the delirium observation scale (DOSS); (minimum score 0 = no delirium; a score of >= 3 means delirium; maximum score 65)
Delirium ICU/MC | up to seven days
  ICU/MC patients' delirium is measured once a day with the Intensive Care Delirium Checklist (ICDSC); (minimum score 0 = no delirium; a score of 1 - 3 means subsyndromal delirium; a score of 4 - 8 means delirium; maximum score 8)
Light | up to six days
  Light level (LUX). This will be measured with a validated application on a mobile phone
Sound | up to six days
  Sound levels (decibel). This will be measured with a validated application on a mobile phone
Hart rate | up to six days
  hart rate is measured with a heart rate monitor and reported every two hours as beats per minute (BPM)
Respiratory rate | up to six days
  Respiratory rate is measured every two hours with a respiratory rate monitor and reported as rate per minute
oxygen saturation | up to six days
  Oxygen saturation is measured every two hours with a oxygen saturation monitor and reported as a percentage
Blood pressure | up to six days
  Blood pressure is measured every two hours with a intra-arterial catheter or a bloodpressure cuff and reported as diastolic value and systolic value (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Bram Tilburgs, Dr., Principal Investigator — adboudumc, intensive care, research

IPD SHARING:
Plan to Share IPD: No